CLINICAL TRIAL: NCT02157675
Title: The Effects of a Polyherbal Supplement on the Signs and Symptoms of Delayed Onset Muscle Soreness: a 2-arm, Randomized, Double-blind, Placebo-controlled, Crossover Design Study
Brief Title: Effects of a Polyherbal Supplement on the Signs and Symptoms of Delayed Onset Muscle Soreness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NewChapter, Inc. (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: NEWC2700; 2013138
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: Delayed onset muscle soreness; Muscle damage; Eccentric exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyherbal capsule (Experimental): Subjects take 1 capsule with breakfast and 1 capsule with lunch. Subjects should take capsules immediately prior to meals and not with carbonated beverages.
  Interventions: Dietary Supplement: Polyherbal capsule
- Placebo capsule (Placebo Comparator): Subjects take 1 capsule with breakfast and 1 capsule with lunch. Subjects should take capsules immediately prior to meals and not with carbonated beverages.
  Interventions: Dietary Supplement: Placebo capsule

INTERVENTIONS:
Dietary Supplement: Polyherbal capsule
  Arms: Polyherbal capsule
Dietary Supplement: Placebo capsule
  Arms: Placebo capsule

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, crossover design study in healthy subjects to determine the effects of a polyherbal supplement on the signs and symptoms of delayed onset muscle soreness (DOMS) induced by eccentric exercise of the arm.

DETAILED DESCRIPTION:
Approximately 30 subjects will be enrolled. The study includes a 19-day treatment period and a minimum 7-day washout period in which no test product is administered. Subjects will then crossover to a second 19-day treatment period to complete the study. Subjects receive test product (polyherbal capsule or placebo capsule) daily during the treatment periods. Two exercise test sessions followed up to 5 days will occur during the study using a modified seated arm-curl bench. Muscle strength is assessed on each day of the 5-day exercise test period. Safety is assessed during the study by collecting adverse events (AEs), clinical laboratory data (serum hematology and chemistry), and vital signs (blood pressure, pulse, respiration rate, temperature).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* be in good general health without clinically significant disease, as determined by medical history, physical examination, and urine drug screens
* body mass index (BMI) ≥ 18 and ≤ 30 kg/m2
* females of child bearing potential must agree to use appropriate birth control methods during the entire study period
* agree not to initiate any new exercise or diet programs during the entire study period
* agree not to change their current diet or exercise program during the entire study period
* understand the study procedures and sign the forms providing informed consent to participate in the study, and authorize the release of relevant protected health information of the study investigator
* agree not to stretch, utilize ice massage, take anti-inflammatory medications (eg, aspirin, ibuprofen), or use any other treatment for the duration of the trial.

Exclusion Criteria:

* previous history of upper extremity injury or pain
* use of anti-inflammatory medications or pain medications beginning at the screening visit and during the study
* daily use of dietary supplements and herbal supplements beginning at the screening visit and during the study
* use of any immunosuppressive drugs or biologic products in the last 12 months (including steroids [except for inhaled and topical dose forms]);
* antibiotic use, anticoagulants, intra-articular steroids in past 3 months
* any significant GI condition that would potentially interfere with the evaluation of the study product including but not limited to inflammatory bowel disease (ulcerative colitis or Crohn's), history of lap band surgery, history of perforation of the stomach or intestines, or gastroparesis
* clinically significant renal, hepatic and biliary, endocrine (including diabetes mellitus), cardiac, pulmonary, pancreatic, neurologic (particularly balance or neuropathy problems), hematologic disorder, or significant mental health disorder
* known allergy or sensitivity to herbal ingredients in the test products, olive oil, or soy
* history or presence of cancer in the last 5 years (except basal cell carcinoma of skin or in-situ cervical cancer)
* recent history of (within 2 years) or strong potential for alcohol or substance abuse
* participation in a clinical study with exposure to any non-registered drug product within 30 days prior to this study
* report use of tobacco or products containing nicotine
* individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk, including subjects who are bed or wheelchair-bound or those who have any physical disability which could interfere with their ability to perform the exercise assessments included in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in peak muscle strength on Day 2 of each test period after eccentric exercise. | Day 2 of each 5-day test period (ie, 48 hours after the eccentric exercise procedure to induce DOMS on Day 0)
  This procedure utilizes 3 sets of 1 repetition of maximal isometric contractions of the arm recorded in pounds and averaged across the 3 sets.

SECONDARY OUTCOMES:
Change from baseline in peak muscle strength after eccentric exercise | Up to 5 days following eccentric exercise.
Change from baseline in pain assessment after eccentric exercise | Days 1-4 of each test period after eccentric exercise
  Pain will be assessed verbally during elbow flexion and extension using a 10-point Likert scale (with 1 = normal, no discomfort and 10 = very uncomfortable).
Change from baseline in flexibility after eccentric exercise | Days 1-4 of each test period after eccentric exercise
  Flexibility of the biceps muscle group will be evaluated with the arm hanging freely at the subject's side. The relaxed extension will be measured using an electronic level and electronic goniometer placed at the elbow.
Change from baseline in elbow girth (swelling) after eccentric exercise | Days 1-4 of each test period after eccentric exercise
  Girth measurements will be taken around the elbow.
Change from baseline in muscle tenderness after eccentric exercise | Days 1-4 of each test period after eccentric exercise
  Muscle tenderness scores will be assessed using a standard manual muscle myometer. Decreasing force application after baseline indicates increasing tenderness, a reflection of muscle damage.
Change from baseline in creatinine kinase (CK) and C-reactive protein (CRP) levels after eccentric exercise | Days 1-4 of each test period after eccentric exercise

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States